CLINICAL TRIAL: NCT00281008
Title: A Phase 2, Double-Blind, Placebo-Controlled, Dose Escalation Study to Assess the Safety, Efficacy, and Pharmacokinetics of ISIS 301012 as Add-on Therapy in Heterozygous Familial Hypercholesterolemia Subjects
Brief Title: Study of ISIS 301012 (Mipomersen) in Heterozygous Familial Hypercholesterolemia Subjects on Lipid Lowering Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012CS9; 2005-004797-24 (EudraCT Number)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Hypercholesterolemia, Familial
Keywords: LDL-cholesterol; apoB-100; Heterozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Cohort A (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort B (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort C (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort D (Experimental): Loading doses followed by extended weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo

INTERVENTIONS:
Drug: ISIS 301012 or Placebo — 50 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, and 36
  Arms: Cohort A
Drug: ISIS 301012 or Placebo — 100 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, and 36
  Arms: Cohort B
Drug: ISIS 301012 or Placebo — 200 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, and 36
  Arms: Cohort C
Drug: ISIS 301012 or Placebo — 300 mg subcutaneous injections on days 1, 4, 8, 11, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, and 85
  Arms: Cohort D

SUMMARY:
The aim of this study is to assess the safety and efficacy of varying doses of ISIS 301012 (mipomersen) as add-on therapy in subjects with Heterozygous Familial Hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 50 kg
* Diagnosis of Heterozygous Familial Hypercholesterolemia.
* Females must be non-pregnant and non-lactating.
* On stable lipid lowering therapy for at least 4 weeks.
* Lipid levels meet the pre-specified criteria.

Exclusion Criteria:

* Subject had heart problems in the prior 6 months.
* Subject has elevated ALT, AST, or CPK.
* History of renal disease, liver disease, or malignancy.
* Use of oral anticoagulants, unless the dose has been stable for 4 weeks
* Have any other conditions, which in the opinion of the Investigator would make the subject unsuitable for enrollment, or could interfere with the subject participating in or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction in LDL-cholesterol from baseline | Week 7 (Cohorts A-C), Week 15 (Cohort D)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (7):
  - Chicago, Illinois
  - Auburn, Maine
  - Scarborough, Maine
  - New York, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Houston, Texas
- Amsterdam, Netherlands